CLINICAL TRIAL: NCT02684032
Title: PHASE 1B STUDY TO ASSESS THE SAFETY, TOLERABILITY, AND CLINICAL ACTIVITY OF GEDATOLISIB IN COMBINATION WITH PALBOCICLIB AND EITHER LETROZOLE OR FULVESTRANT IN WOMEN WITH METASTATIC OR LOCALLY ADVANCED/RECURRENT BREAST CANCER (MBC)
Brief Title: A Study To Assess The Tolerability And Clinical Activity Of Gedatolisib In Combination With Palbociclib/Letrozole Or Palbociclib/Fulvestrant In Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celcuity Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2151009
Record Dates: First submitted 2016-02-10; First posted 2016-02-17 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: PI3K (phosphoinositide 3-kinase); mTOR (mechanistic target of rapamycin); PI3K/mTOR; metastatic breast cancer (MBC); ER+ (estrogen receptor positive); HER2- (human epidermal growth factor receptor 2 negative)
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — gedatolisib; palbociclib; Letrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Letrozole Cohort (Experimental): Letrozole combination cohort in dose escalation
  Interventions: Drug: Gedatolisib; Drug: Palbociclib; Drug: Letrozole
- Fulvestrant cohort (Experimental): Fulvestrant combination cohort in dose escalation
  Interventions: Drug: Gedatolisib; Drug: Palbociclib; Drug: Fulvestrant
- ARM A (Experimental): Gedatolisib + palbociclib + letrozole in dose expansion
  Interventions: Drug: Gedatolisib; Drug: Palbociclib; Drug: Letrozole
- ARM B (Experimental): Gedatolisib + palbociclib + fulvestrant in dose expansion
  Interventions: Drug: Gedatolisib; Drug: Palbociclib; Drug: Fulvestrant
- ARM C (Experimental): Gedatolisib + palbociclib + fulvestrant in dose expansion
  Interventions: Drug: Gedatolisib; Drug: Palbociclib; Drug: Fulvestrant
- Arm D (Experimental): Gedatolisib (3:1) + palbociclib + fulvestrant in dose expansion
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Gedatolisib — Gedatolisib weekly intravenous starting at 180 mg/week in a 4 week cycle.
  Arms: ARM A; ARM B; ARM C; Fulvestrant cohort; Letrozole Cohort
Drug: Palbociclib — Palbociclib initiated at 125 mg daily: 3 out of 4 weeks in a 4 week cycle.
  Arms: ARM A; ARM B; ARM C; Fulvestrant cohort; Letrozole Cohort
Drug: Letrozole — Letrozole at 2.5 mg daily
  Arms: ARM A; Letrozole Cohort
Drug: Fulvestrant — Fulvestrant administered intramuscularly at 500 mg on Day 1, 15 and 28 and then every 28 days.
  Arms: ARM B; ARM C; Arm D; Fulvestrant cohort

SUMMARY:
This is a multicenter, open label, Phase 1b study in patients with mBC. This study will have a dose escalation to identify the maximum tolerated dose (MTD) of the combination of gedatolisib plus palbociclib/fulvestrant and gedatolisib plus palbociclib/letrozole and expansion to estimate the objective response rate (OR) of the combination of gedatolisib plus palbociclib/letrozole or palbociclib/fulvestrant.

DETAILED DESCRIPTION:
This is a multicenter, open label, continuous Phase 1b study in patients with MBC. This study will have a dose escalation and expansion. The dose escalation will identify the maximum tolerated dose (MTD) of the combination of gedatolisib plus palbociclib/fulvestrant and gedatolisib plus palbociclib/letrozole. The expansion will estimate the objective response rate (OR) of the combination of gedatolisib plus palbociclib/letrozole and the combination of gedatolisib plus palbociclib/fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older, who are either: Postmenopausal or Pre/perimenopausal women with medically-induced menopause by treatment with agents to induce chemical menopause.
* Histologically or cytologically proven diagnosis of breast cancer with evidence of metastasis.
* Documentation of estrogen receptor positive ((ER+), human epidermal growth factor receptor 2 (HER2 negative (HER2-)) tumor.
* Dose Escalation Portion: Patients must satisfy one of the following criteria:

  * Letrozole combination cohort (L): metastatic breast cancer (MBC) with progression who are candidates for a letrozole-containing regimen, with palbociclib.
  * Fulvestrant combination cohort (F): MBC with progression who are candidates for a fulvestrant containing regimen, with palbociclib.
* Dose Expansion Portion: Patients must satisfy one of the following criteria:

  * Arm A: MBC with progression and no prior endocrine based systemic therapy in the metastatic setting;
  * Arm B: MBC with progression during or following one prior endocrine based systemic therapy in the metastatic setting, with no prior therapy with any cyclin-dependent kinase (CDK) inhibitor;
  * Arm C/Arm D: MBC with progression during or following one or two prior endocrine based systemic therapies in the metastatic setting, and following prior therapy with a CDK inhibitor.
* Measurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
* Bone only patients during dose escalation portion.
* Availability of archival tumor biopsy sample or willing to provide fresh biopsy if not available.
* Eastern Cooperative Oncology Group [ECOG] performance must be 0 or 1.
* Adequate bone marrow, renal and liver function.

Exclusion Criteria:

* Prior treatment with a mechanistic target of rapamycin (mTOR) inhibitor or phosphoinositide 3-kinase (PI3K) inhibitor.
* More than 1 line of prior chemotherapy in the treatment of metastatic or locally advanced/recurrent disease.
* Bone only patients during expansion/efficacy portion.
* Patients with advanced/metastatic disease who have symptomatic visceral spread, and who have life threatening complications needing immediate therapy, such as massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver replacement with tumor.
* Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases.
* Active bacterial, fungal or viral infection.
* Uncontrolled or significant cardiovascular disease.
* Radiation therapy within 4 weeks of investigational product.
* Cytotoxic chemotherapy within 4 weeks of investigational product (6 weeks for mitomycin C or nitrosoureas) if immediate prior regimen was administered on an every 3 4 week schedule or 2 weeks of investigational product if immediate prior regimen consisted of weekly therapy.
* Any other anti cancer agents (eg, hormonal, biological, investigational) within 5 times the half life prior to investigational product.
* Impairment of gastro intestinal (GI) function or GI disease.
* Pregnant female patients; breastfeeding female patients; and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study and for 90 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 141 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | up to 28 days
Objective response rate observed in patients in the dose expansion portion | 16 weeks
  Number of patients for each response category, objective response rate (number of patients with a complete response (CR)) relative to the number of response evaluable patients
Objective response rate observed in patients in the dose expansion portion | 16 weeks
  Number of patients for each response category, objective response rate (number of patients with a partial response (PR)) relative to the number of response evaluable patients)

SECONDARY OUTCOMES:
Tumor response observed in patients in the dose escalation portion | 16 weeks
Duration of response | 16 weeks
QTc interval (corrected QT interval) | Screening up to 6 months
  The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle.
Maximum observed plasma concentration | Day 1: 0, 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 24, 72 and 168 hours. Cycle 2 Day 1: 0, 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 24, 72 and 168 hours
Progression free survival | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Igor Gorbatchevsky, MD, Study Director — Celcuity Inc
Locations (39):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Compassionate Care Research Group Inc. at Compassionate Cancer Care Medical Group, Inc., Corona, California
  - Compassionate Care Research Group Inc. at Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Keck Hospital of USC - Norris Healthcare Center (HC3), Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center / Investigational Drug Services, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Compassionate Care Research Group Inc. at Compassionate Cancer Care Medical Group, Inc., Riverside, California
  - UCSF - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AiP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - University of Colorado Hospital - Clinical Trials Office (CTO), Aurora, Colorado
  - University of Colorado Hospital- Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Moffitt Cancer Center Richard M Schulze Family Foundation Outpatient Center at McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - UNC Cancer Hospital Infusion Pharmacy, Chapel Hill, North Carolina
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Ohio State University Wexner Medical Center James Cancer Hospital, Columbus, Ohio
  - Stefanie Spielman Comprehensive Breast Cancer, Columbus, Ohio
  - Thomas Jefferson University - Clinical and Regulatory, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - U.T. MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Seattle Cancer Care Alliance (SCCA) Investigational Drug Services, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Celcuity will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.

REFERENCES:
- [Derived] Layman RM, Han HS, Rugo HS, Stringer-Reasor EM, Specht JM, Dees EC, Kabos P, Suzuki S, Mutka SC, Sullivan BF, Gorbatchevsky I, Wesolowski R. Gedatolisib in combination with palbociclib and endocrine therapy in women with hormone receptor-positive, HER2-negative advanced breast cancer: results from the dose expansion groups of an open-label, phase 1b study. Lancet Oncol. 2024 Apr;25(4):474-487. doi: 10.1016/S1470-2045(24)00034-2. PMID 38547892
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B2151009